CLINICAL TRIAL: NCT04599114
Title: Virtual for Care Atrial Fibrillation Patients Using VIRTUES (Virtual Integrated Reliable Transformative User-Driven E-Health System)
Brief Title: Virtual for Care Atrial Fibrillation Patients Using VIRTUES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other)
Responsible Party: Principal Investigator, Allan Skanes, Director, Electrophysiology Laboratory, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4411
Record Dates: First submitted 2020-10-02; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation
Keywords: Virtual care
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study will use a retrospective chart review to examine characteristics of patients who present to the emergency room with atrial fibrillation as well as a non-randomized prospective cohort who will be offered enrollment into the virtual platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIRTUES Arm (Experimental): Patients in the VIRTUES arm will be offered enrollment into the virtual atrial fibrillation care platform.
  Interventions: Behavioral: VIRTUES

INTERVENTIONS:
Behavioral: VIRTUES — VIRTUES is a digital health platform that offers 2 way communication between clinicians and patients to address symptoms stemming from atrial fibrillation.

SUMMARY:
Patients will atrial fibrillation, a type of irregular heart rhythm, frequently go to the emergency room in order to manage their condition. This study will use a chart review to look at the characteristics and frequency of atrial fibrillation patients who go to the emergency room. In addition to the chart review, patients with atrial fibrillation who have recently gone to the emergency room or have been hospitalized will be approached and asked if they want to use an electronic health care system that can be accessed by both themselves and their health care providers. Along with the system, patients will be given a Health Canada approved heart rhythm sensor, so patients will be able to record their heart rhythm when they feel symptoms and send the information to the heart rhythm team. The heart rhythm team will then make real-time recommendations to the patient about how they can manage their rhythm and symptoms. Patients will be asked to complete satisfaction and quality of life surveys. Our goal is to provide efficient and effective care for patients with AF, resulting in decreased repeat ED visits.

DETAILED DESCRIPTION:
See brief summary.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* documented symptomatic new-onset or pre-existing, non-valvular AF
* ER visit or hospitalization for primary AF in the last 6 months
* proficient in the English language

Exclusion Criteria:

* unable to provide informed consent
* planning to move/relocate during the period of study
* current pregnancy
* patient is a prisoner/incarcerated
* no access to a smart device with Bluetooth capabilities
* planned percutaneous coronary intervention, coronary artery bypass graphing or heart valve surgery within the next year
* any medical condition making 1 year survival unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who present to the emergency department due to atrial fibrillation, after their index visit | 12 months
  See title

SECONDARY OUTCOMES:
Number of AF-related ER visit per patient, post index visit | 12 months
  See title
Utility of the system | 12 months
  Number of uses of the system/patient, number of accesses to the health record, number of heart rhythm VIRTUES team - patient feedbacks on the VIRTUES app, percentage of care plans followed by the patient
Survey-based experience with the VIRTUES application | Baseline, 3 months, 12 months
  Survey-based experience will be determined by the "Virtual AF Care Patient Satisfaction Questionnaire". The questionnaire consists of 5 questions regarding the VIRTUES platform using a 5 point likert scale (strongly agree to strongly disagree) in addition to a final open ended question asking for feedback regarding the application.
Pre and post patient reported outcomes using the Atrial Fibrillation Effect on Quality of Life (AFEQT) Questionnaire and the EQ-5D-5L | Baseline, 3 months, 12 months
  The Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) questionnaire is a well-validated questionnaire with 2 sections. The first section asked about a patient's incidence of atrial fibrillation, the second section inquires as to the presence of atrial fibrillation symptomsand how limiting they were. In general, higher scores mean more frequent atrial fibrillation symptoms that are very/extremely limiting and bothersome.
Time to stroke/TIA, systematic embolism, cardiovascular (CV) hospitalization, death | 12 months
  The length of time between index presentation for atrial fibrillation and the onset of any of the above conditions will be calculated for both the retrospective and prospective cohorts.
Frequency of stroke/TIA, systematic embolism, cardiovascular (CV) hospitalization, death | 12 months
  The number of any of the above conditions occurring in both the retrospective and prospective cohorts will be counted and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Allan C Skanes, Md, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (3):
- Canada (3):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Rachel Caris, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No